CLINICAL TRIAL: NCT06665139
Title: The Relationship Between the Thickness of the Muscles Stabilizing the Scapula and Pain in Impingement Syndrome
Brief Title: the Thickness of the Muscles and Pain in Impingement Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cansin Medin, Principle investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2024/50
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Impingement Shoulder; Impingement Syndrome; Pain, Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- impigment: Patients diagnosed with impingement and meeting the criteria will be included,
  Interventions: Diagnostic Test: muscle thickness
- healty: the healthy group will consist of hospital staff who do not have shoulder pain and who are not diagnosed with a shoulder-related disease.
  Interventions: Diagnostic Test: muscle thickness

INTERVENTIONS:
Diagnostic Test: muscle thickness — Pain intensity will be measured with visual analog scale, sonographic severity grade of shoulder impingement syndrome, muscle thickness of serratus anterior muscle, upper trapezius and middle trapezius with USG in patients diagnosed with impingement and meeting the criteria and healthy volunteers.

SUMMARY:
Pain intensity will be measured with visual analog scale. Sonographic severity grade of shoulder impingement syndrome, serratus anterior muscle, upper trapezius and middle trapezius will be measured with USG in patients diagnosed with impingement and meeting the criteria and healthy volunteers.

DETAILED DESCRIPTION:
Patients diagnosed with impingement and meeting the criteria will be included, while the healthy group will consist of hospital staff who do not have shoulder pain and who are not diagnosed with a shoulder-related disease. Pain intensity will be measured with VAS (visual analog scale), the sonographic severity grade of shoulder impingement syndrome, the serratus anterior muscle, the upper trapezius and the middle trapezius will be measured with USG.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Cognitive ability to understand test instructions
* Symptom duration longer than 1 month
* At least two positive Neer, Hawkins and painful arch tests

for healty volunteers

* 18-65 years
* cognitive ability to understand test instructions
* negative impingment test

Exclusion Criteria:

* Fibromyalgia
* cervical radiculopathy
* those who have received injections or physical therapy in the last month
* Those with a disorder that may affect shoulder joint range of motion and muscle mass (previous fracture, surgery, subluxation)
* BMI over 35
* inflammatory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with impingement and meeting the criteria will be included, while the healthy group will consist of hospital staff who do not have shoulder pain and who are not diagnosed with a shoulder-related disease.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
sonographic severity grade of shoulder impingment syndrome | baseline
  The distance between the acromion and the greater tuberosity will be measured in both neutral and dynamic positions, and the disease severity will be assessed according to the ratio between these two data.

CONTACTS AND LOCATIONS:
Overall Officials: cansın medin ceylan, MD, Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Cansın Medin Ceylan, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No